CLINICAL TRIAL: NCT07025447
Title: Cluster-Randomized Controlled Trial of a Father-Inclusive Parenting Intervention in Mwanza, Tanzania
Brief Title: Father-Inclusive Parenting Intervention in Mwanza, Tanzania
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Tanzania Home Economics Organization (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Joshua Jeong, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00006498; 5R00HD105984 (NIH)
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Parents
Keywords: Fatherhood; Parenting; Caregiving; Early childhood development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Familia Bora (Experimental): Participants will be offered a parenting group program available in their community, with weekly scheduled sessions for approximately 5 months.
  Interventions: Behavioral: Familia Bora
- Control Group (No Intervention): Participants will not receive any intervention.

INTERVENTIONS:
Behavioral: Familia Bora — Familia Bora is a couples-based group parenting program that takes place in a preferred location within the community among participants. Twelve couples will be enrolled in each village and form one parenting group. CHWs will be trained to deliver the intervention.
  The program will involve 17 group sessions. Each session is expected to last 1.5 hours and will be delivered weekly for approximately 5 months. Each session will focus on various topics, including responsive caregiving, positive discipline, managing emotions and stress management, child nutrition, couples' communication, non-violent conflict resolution strategies in relationships, gender equity, and early child care and education. In addition to the weekly group parenting sessions, CHWs will be encouraged to conduct home visits to engage couples who miss sessions, reinforce key messages, and provide extra support for caregivers and children as needed.
  Arms: Familia Bora

SUMMARY:
This cluster-randomized controlled trial aims to evaluate the impact of a couples-based parenting program, "Familia Bora," on mothers' and fathers' parenting, couples' relationships, gender, and early child development in the Mwanza Region, Tanzania. Additionally, this study aims to assess the program's implementation and identify factors influencing its quality and effectiveness.

Trained community health workers will deliver the program by facilitating weekly peer group sessions in their villages. Twelve couples with a child under two years old will be enrolled in each village. The program will cover various topics, including responsive caregiving, positive discipline, stress management, healthy couples' communication, nutrition, and gender.

DETAILED DESCRIPTION:
An estimated 43% of children under five in low- and middle-income countries are at risk of not achieving their developmental potential, with the burden highest in sub-Saharan Africa. While there is robust evidence on the effectiveness of parenting interventions for improving nurturing care and early childhood development (ECD), the vast majority of existing programs have targeted mothers exclusively. Fathers are often excluded from parenting programs, even though evidence highlights their vital contributions to child and family wellbeing.

This cluster-randomized controlled trial will evaluate the impacts and implementation quality of a newly developed, culturally-responsive, gender-transformative, and father-inclusive parenting intervention ("Familia Bora"). The study will be implemented in 33 villages across Misungwi and Sengerema districts in Mwanza Region, Tanzania. Half of the villages will be randomly assigned to the intervention (17 villages) versus control group (16 villages) with stratification by district. The program will train community health workers (CHWs) to deliver the program to groups of 12 randomly selected couples per village.

Familia Bora primarily involves group sessions covering various topics, including responsive parenting, positive discipline, couples' communication, stress management, and gender roles in family caregiving. These group sessions will be held at a convenient community location on a weekly basis for approximately five months.

In total, the trial will enroll 396 couples with young children (i.e., 396 men and 396 female partners). Quantitative surveys will be conducted with fathers and mothers at baseline and endline to assess outcomes, including maternal and paternal parenting practices and attitudes, gender attitudes, relationship dynamics, and early childhood development. Quantitative data will be collected from CHWs at baseline and endline to assess program-related changes in their knowledge, attitudes, and skills. In addition to the quantitative evaluation, qualitative methods will be used to evaluate implementation processes and participant perspectives through midline and endline in-depth interviews with a subsample of caregivers and CHWs, community leaders, and other relevant stakeholders across the intervention villages.

ELIGIBILITY:
Eligibility criteria for couples:

Inclusion Criteria:

* Each individual is an adult aged 18-65 years
* Each individual is the primary female or male caregiver of a child younger than 2 years of age
* The two individuals are currently in a marital or partnered relationship with each other
* Both individuals have lived in the same household as each other and the child during the past month, and
* Both individuals provide written informed consent to participate in the study.

Exclusion Criteria:

* Need to satisfy the inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 792 (Actual)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Parental stimulation score | Baseline, 6 months
  Maternal and paternal stimulation practices will be measured by the Family Care Indicators (FCI), which are reported in terms of the number of developmentally-enriching activities that the parent engaged with the young child in the past week (e.g., singing, telling stories). Activities adapted from the Family Care Indicators. The total score ranges from 0 to 7, with higher scores indicating greater parental engagement in stimulation activities.

SECONDARY OUTCOMES:
Caregiver Reported Early Development Instrument (CREDI) long form | Baseline, 6 months
  Early child development will be measured using the Caregiver Reported Early Development Instrument (CREDI) long form. It relies on parental reporting and assesses four domains of early developmental milestones: motor, language, cognitive, and socioemotional development. Higher scores reflect a greater number of age-appropriate developmental skills as reported by caregivers.
Variety of early learning materials score | Baseline, 6 months
  Play and learning materials will be measured using the Early Childhood Development Module of the Multiple Indicator Cluster Survey. Includes types of different objects children play with at home (e.g., homemade toys, manufactured toys, household objects) as well as the number of books present in the household. Play and learning modules will be reported by the mother.
Parental disciplinary practices score | Baseline, 6 months
  Maternal and paternal disciplinary practices will be reported in terms of harsh punishment (e.g., shook the child, shouted at the child) and positive disciplinary practices (e.g., explained why the behavior was wrong) used by the parent towards the child. Items were adapted from the Child Discipline Module of the Multiple Indicator Cluster Survey, with additional items related to verbal harsh punishment and positive reinforcement created by the study team based on formative research within this study context. Separate indicators will be created for the use of any harsh disciplinary practices or any positive disciplinary practices. Higher values on each indicator will reflect greater use of the respective disciplinary practice (i.e., harsh or positive).
Level of father involvement in childcare and household chores | Baseline, 6 months
  The level of the fathers' involvement will be self-reported by men as well as through maternal reports about their male partners regarding the number of childcare and household activities performed by the father to support the young child, female partner, and family more broadly (e.g., bathing the child, providing money to the partner, washing dishes/clothes). Measure developed and validated by the authors. Higher scores indicate greater fathers' involvement in childcare activities and household chores.
Parenting attitudes score | Baseline, 6 months
  Attitudes toward parenting will be reported by mothers and fathers using a tool developed by the study team, informed by formative qualitative research conducted in the study context. The tool captures agreement with statements related to developmentally appropriate parenting, general parenting practices, and discipline approaches. Higher scores reflect more positive attitudes toward parenting.
Gender attitudes score | Baseline, 6 months
  Gender attitudes reported by mothers and fathers regarding gender norms around childcare and domestic responsibilities, household equity, and power dynamics within partner relationships. This measure was developed by the study team based on formative research in this context. Higher scores indicate more gender-equitable attitudes
Decision-making score | Baseline, 6 months
  Mothers and fathers will report on who in their family (mother, father, someone else, or shared) has the final say about decisions across various family domains. Items were adapted from the decision-making module of the Demographic Health Surveys. Women's decision-making autonomy will be scored as the number of domains in which she is involved, with higher scores indicating greater participation.
Parenting stress score | Baseline, 6 months
  Parenting distress will be reported by mothers and fathers using the Parenting Stress Index-Short Form, Parental Distress subscale. The scale is based on a series of statements that parents can agree or disagree with, and the scores are calculated by summing the responses to the items. Higher scores indicate greater levels of stress.
Maternal intimate partner violence victimization | Baseline, 6 months
  Mothers will report on their experiences of intimate partner violence in the past three months using a standardized set of violent acts perpetrated by their partner (i.e., the child's father), adapted from the World Health Organization's multi-country study on women's health and domestic violence against women. The primary IPV indicator will be a proportion reflecting the percentage of mothers who report experiencing any form of IPV. In addition, we will calculate separate binary indicators for each type of IPV (physical, sexual, and emotional).
Child dietary diversity | Baseline, 6 months
  Child dietary diversity will be reported by mothers as the number of food groups (out of eight) consumed by the child in the previous 24 hours, following World Health Organization (WHO) guidelines. This measure is assessed in children aged six months and older, with higher scores indicating a greater likelihood of achieving a nutritionally adequate diet.

OTHER OUTCOMES:
Child epigenetic pace of aging | 6 months
  Methylation pace of aging was developed from DNA-methylation analysis of Pace of Aging in the Dunedin Study birth cohort (DunedinPACE). Pace of Aging is a composite phenotype derived from analysis of longitudinal change in 18 biomarkers of organ-system integrity (Belsky et al., 2015). Increments of methylation pace of aging correspond to "years" of physiological change occurring per 12-months of chronological time.
Child DNA methylation | 6 months
  Salivary DNA-methylation profiles of cognitive functioning, i.e., "Epigenetic-g", can be computed on the basis of weights from a blood-based epigenome wide association study of general cognitive functions (g) in adults. General cognitive ability was derived from the first unrotated principal component of logical memory, verbal fluency and digit symbol tests, and vocabulary. Epigenetic-g is conceptually distinct from biological aging. If a higher quality measure of epigenetic profile of cognitive functioning becomes available at the time of analysis, we will substitute that instead.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Jeong, ScD, Principal Investigator — Emory University
Locations (2):
- Emory University, Atlanta, Georgia, United States
- Communities in Mwanza,Tanzania, Mwanza, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
The investigator will share de-identified Individual participant data that underlie the results reported in the primary trial article.
Supporting Information: Study Protocol
Time Frame: Data will be shared beginning 6 months and ending 36 months following article publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal to achieve the aims in the approved proposal.
  Proposals should be directed to Joshua.jeong@emory.edu. To gain access, data requestors will need to sign a data access agreement.